CLINICAL TRIAL: NCT04216030
Title: Iron Bioavailability From Iron Bio-fortified Irish Potato in Peruvian Women Between 18-25 Years of Age.
Brief Title: IP Peru, Bioavailability of Iron From Potatoes
Acronym: IPPERU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: Genetics, Genomics and Crop Improvement Program, International Potato Center, Lima, Peru (Unknown); United States Agency for International Development (USAID) (U.S. Federal Agency); Quadram Institute Bioscience (Other); Instituto de Investigacion Nutricional, Lima, Peru (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 1267-USAI-000-ETH-01
Record Dates: First submitted 2019-12-29; First posted 2020-01-02 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Iron-deficiency; Iron Deficiency Anemia; Iron Deficiency (Without Anemia)
Keywords: Biofortification; Staple crops; Stable isotope studies
MeSH Terms: conditions — Anemia, Iron-Deficiency; Iron Deficiencies

STUDY DESIGN:
Intervention Model Description: Each woman consumes both high-iron Irish potato and a regular Irish potato variety.
Masking Description: Participant is non-blinded based on differences in meal option A and B, meal option A --> B or B --> A, is assigned through investigator randomisation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High iron Irish potato (Experimental): Meal sequence B, IP High Fe
  Interventions: Other: High Fe IP meal labelled with Fe-58
- Regular Irish potato (Active Comparator): Meal sequence A, OFSP control
  Interventions: Other: Control OFSP meal labelled with Fe-57

INTERVENTIONS:
Other: High Fe IP meal labelled with Fe-58 — 500 gram steamed, mashed OFSP high Fe with 0.33 mg FeSO4-58 daily for 10 days
  Arms: High iron Irish potato
Other: Control OFSP meal labelled with Fe-57 — 500 gram steamed, mashed OFSP control with 0.33 mg FeSO5-57 daily for 10 days
  Arms: Regular Irish potato

SUMMARY:
To combat iron deficiency in Low and Middle-Income Countries, sustainable food-based solutions have to be implemented to serve populations, not only individuals. One solution is the introduction of iron biofortified staple crops on market level. Before market level introduction, the bioavailability of iron in the new biofortified Irish Potato (IP) breed needs to be assessed. In this study the investigator compares the fractional and total iron absorption after extrinsic stable isotope labelling of the new biofortified high iron IP variety and a normal market level IP variety. The study is conducted in Peruvian women of reproductive age with marginal iron status.

DETAILED DESCRIPTION:
The 40 women enrolled will consume test meals consisting of 500g steamed and mashed high iron Irish potatoes labelled with Fe-58 daily for a period of 10 days and will then switch to the test meals consisting of 400g steamed and mashed control sweet potatoes labelled with Fe-57 for a period of 10 days. The order of test meal type is random. A baseline blood sample will be taken on the first meal feeding day prior to consumption of any test meals, study day 15 (before switching to the other test meal IP variety), on study day 26 (14 days after completion of the first test meal period) and on Day 40 (14 days after completion of the second test meal period). Erythrocyte incorporation of the stable isotope labels will be measured in these blood samples using an ICPMS and will be used to calculate fractional and total iron absorption from the two different type of test meals.

ELIGIBILITY:
Inclusion Criteria:

1. Woman aged 18-25 years old.
2. Low/marginal iron status: serum ferritin (SF) ≤ 25 μg/L.
3. Normal BMI for age (18.5-25.0 kg/m2).
4. Weight less than 65 kg. We will give equal amounts of stable isotopes to each study participant and therefore need to set a limit on body weight in order to achieve measurable isotope enrichment in erythrocytes.
5. Willing and able to commute to the meal distribution/health centre site.
6. Able to understand and to sign written concept prior to trial entry.
7. Informed consent signed.
8. Prepared to use contraceptives for the duration of the study

Exclusion Criteria:

1. Severe anaemia Hb <107.2 g/L (adjusted for meters above sea level)
2. Inflammation/infection (CRP > 5 mg/100 ml).
3. Relevant digestive (intestinal, gastric, hepatic or pancreatic), renal, metabolic disease, and any other problem that will interfere with the study as determined by the screening visit and by self-report from the subjects.
4. Pregnant (urine test before entering the study) or breast-feeding.
5. Any medication or supplement which may impact iron metabolism.
6. Unwilling to discontinue vitamin and minerals supplements at least two weeks prior to the study start, as ascertained at the screening visit.
7. Significant blood losses over the past 6 months (i.e. trauma, major surgery, blood donation).
8. Subject who cannot be expected to comply with study procedures.
9. Presence of fever (>37.5 °C) on the first study day

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2019-05-14 (Actual); Primary Completion 2019-08-08 (Actual); Study Completion 2019-08-08 (Actual)

PRIMARY OUTCOMES:
Fractional iron absorption from both Irish Potato test meals | Measured 2 weeks after completion of feeding day sequence. Sequence consist of 2 times 10 feeding days.
  Proportion of stable isotope administered with test meals that has been incorporate into erythrocytes 14 days after completion of specific test meal feeding period
Total iron absorption from both Irish Potato test meals | Measured 2 weeks after completion of feeding day sequence. Sequence consist of 2 times 10 feeding days.
  Amount of iron absorbed (mg) from the labelled test meals

SECONDARY OUTCOMES:
Concentration of plasma ferritin level | screening (-1), day 1 (baseline), day 15 (before switch to other test meal type) day 26 (last feeding day) and day 40 (14 days after last test meal consumption).
  Iron status marker
Concentration of plasma CRP level | screening (-1), day 1 (baseline), day 15 (before switch to other test meal type) day 26 (last feeding day) and day 40 (14 days after last test meal consumption).
  Inflammation status marker

CONTACTS AND LOCATIONS:
Overall Officials: Reyna Liria, Principal Investigator — INN; Mary Penny, Principal Investigator — INN
Locations (1):
- Instituto de Investigacion Nutricional, Lima, Peru

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jongstra R, Mwangi MN, Burgos G, Zeder C, Low JW, Mzembe G, Liria R, Penny M, Andrade MI, Fairweather-Tait S, Zum Felde T, Campos H, Phiri KS, Zimmermann MB, Wegmuller R. Iron Absorption from Iron-Biofortified Sweetpotato Is Higher Than Regular Sweetpotato in Malawian Women while Iron Absorption from Regular and Iron-Biofortified Potatoes Is High in Peruvian Women. J Nutr. 2020 Dec 10;150(12):3094-3102. doi: 10.1093/jn/nxaa267. PMID 33188398